CLINICAL TRIAL: NCT06217367
Title: Do Common Over-the-counter Antihistamine Medications Modify Thermoregulatory Responses During Passive Heat Stress?
Brief Title: Over-the-Counter Antihistamines & Heat Stress
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Nicholas Ravanelli, Principal Investigator, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 100241; 273752 (Registry Identifier: Health Canada, Control Number)
Record Dates: First submitted 2023-11-08; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Heat Illness; Allergic Rhinitis; Heat Injury; Sudomotor Sympathetic Dysfunction
Keywords: H1 antihistamine; Sweating; Heat stress; Thermoregulation; M3 Muscarinic receptors; H1 receptor antagonism; M3 Muscarinic receptor blockade; Heat Illness/Injury; Allergic Rhinitis; Over-the-counter antihistamines; Allergy medication
MeSH Terms: conditions — Heat Stress Disorders; Rhinitis, Allergic; Wounds and Injuries; Drug Hypersensitivity | interventions — Diphenhydramine; Loratadine; desloratadine; Sugars

STUDY DESIGN:
Intervention Model Description: Each participant will be asked to ingest either i) 50mg of diphenhydramine, ii) 10 mg loratadine iii) 5 mg desloratadine, or iv) placebo (sugar pill) ~2 hours before heating protocol in a random pre-determined order over four separate experimental trials.
Who Masked: Participant, Investigator
Masking Description: Participants will be informed of the study interventions prior to experimental trials to ensure participants are able to provide informed consent. However, participants will blinded to the order of the arms (i.e., participants will not be informed which antihistamine/placebo pill they ingest for any trial). Data will remain blinded to researchers until after a third-party statistical analysis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 50 mg Diphenhydramine (Experimental)
  Interventions: Drug: 50 mg Diphenhydramine
- 10 mg Loratadine (Experimental)
  Interventions: Drug: 10 mg Loratadine
- 5 mg Desloratadine (Experimental)
  Interventions: Drug: 5 mg Desloratadine
- Placebo (Sugar pill) (Placebo Comparator)
  Interventions: Other: Placebo (Sugar Pill)

INTERVENTIONS:
Drug: 50 mg Diphenhydramine — Participants ingest 50mg of diphenhydramine orally ~2 hours prior to a passive heating protocol. Participants then don a water-perfusion heat suited and lay supine on assessment table while 49℃ is circulated throughout the garment. Heating persists until participants reach a 1.5℃ increase in core temperature from baseline.
  Other Names: Benadryl®
  Arms: 50 mg Diphenhydramine
Drug: 10 mg Loratadine — Participants ingest 10 mg of loratadine orally ~2 hours prior to a passive heating protocol. Participants then don a water-perfusion heat suited and lay supine on assessment table while 49℃ is circulated throughout the garment. Heating persists until participants reach a 1.5℃ increase in core temperature from baseline.
  Other Names: Claritin®
  Arms: 10 mg Loratadine
Drug: 5 mg Desloratadine — Participants ingest 5 mg of desloratadine orally ~2 hours prior to a passive heating protocol. Participants then don a water-perfusion heat suited and lay supine on assessment table while 49℃ is circulated throughout the garment. Heating persists until participants reach a 1.5℃ increase in core temperature from baseline.
  Other Names: Aerius®
  Arms: 5 mg Desloratadine
Other: Placebo (Sugar Pill) — Participants ingest placebo pill orally ~2 hours prior to a passive heating protocol. Participants then don a water-perfusion heat suited and lay supine on assessment table while 49℃ is circulated throughout the garment. Heating persists until participants reach a 1.5℃ increase in core temperature from baseline.
  Arms: Placebo (Sugar pill)

SUMMARY:
Allergic rhinitis (AR) currently affects ~25% of Canadians, and due to factors of climate change, this number is expected to increase over the coming decade. AR symptoms can significantly impact individuals' quality of life by compromising sleep, productivity, and social interactions. To alleviate AR symptoms, North Americans tend to rely on H1 antihistamine medications available over-the-counter (OTC) at most pharmacies. However, public health authorities currently suggest restraining all antihistamines during heat waves due to beliefs that M3 muscarinic receptor and H1 receptor antagonism, independent pharmacological mechanisms of H1 antihistamines, might suppress thermoregulatory responses to heat stress and increase individuals' susceptibility to heat-related illness/injury. To date, studies using supramaximal doses of antihistamines have demonstrated reductions in sweating, however these doses and administration routes are not the typical use case. Additional studies utilizing fexofenadine, a second-generation H1 antihistamine, have linked H1 receptor antagonism to reductions in skin blood flow, potentially impacting thermoregulation by reducing peripheral blood redistribution. Empirical evidence supporting OTC H1 antihistamines impacting thermoregulatory control at recommended doses is scarce. Thus, this study aims to systematically assess whether three common OTC H1 antihistamines, taken as prescribed, alter thermoregulatory responses during thermal stress.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between ages 19 and 39 years
* Fully vaccinated against COVID-19
* Able to provide informed consent
* Body-mass index under 30

Exclusion Criteria:

* Body-mass index over 30
* Currently taking sedative or autonomic nervous system depressant medication
* Hypersensitivity to diphenhydramine, loratadine, or desloratadine
* History of cardiovascular disease, cancer, type 1 or 2 diabetes, chronic obstructive pulmonary disorder, or cystic fibrosis
* Have smoked tobacco products less than 12 months prior to participation
* Pregnant/Breastfeeding

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Whole-Body Sweat Losses | For each study arm (all completed within 4 months), measurements taken immediately before heating protocol & immediately following the heating protocol
  Difference in participants' pre/post body mass
Skin Blood Flow | For each study arm (all completed within 4 months), measured before heating, and at every 0.25C increase in core temperature (+0.25C, +0.50C, +0.75C, +1.0C, +1.25C, and +1.5C), or every ~15 minutes of (up to ~90 minutes) and immediately after heating
  Measured using laser-doppler skin blood blow sensor affixed to forearm
Heart Rate | For each study arm (all completed within 4 months), measured before heating, and at every 0.25C increase in core temperature (+0.25C, +0.50C, +0.75C, +1.0C, +1.25C, and +1.5C), or every ~15 minutes of (up to ~90 minutes) and immediately after heating
  Measured using electrocardiogram
Mean Arterial Pressure | For each study arm (all completed within 4 months), measurements taken at baseline before heating, and every 10 minutes throughout heating protocol (up to ~ 90 minutes), and immediately after heating
  Measured using brachial blood pressure cuff
Local Sweat Rate | For each study arm (all completed within 4 months), measured before heating, and at every 0.25C increase in core temperature (+0.25C, +0.50C, +0.75C, +1.0C, +1.25C, and +1.5C), or every ~15 minutes of (up to ~90 minutes) and immediately after heating
  Measured using ventilated sweat capsules affixed to forearm and chest

SECONDARY OUTCOMES:
Thermal Sensation | For each study arm (all completed within 4 months), measured before heating, and at every 0.25C increase in core temperature (+0.25C, +0.50C, +0.75C, +1.0C, +1.25C, and +1.5C), or every ~15 minutes of (up to ~90 minutes) and immediately after heating
  Self-assessments of thermal sensation using a 7-point analog scale where -3 is "Cold" and +3 is "Hot".
Thermal Comfort | For each study arm (all completed within 4 months), measured before heating, and at every 0.25C increase in core temperature (+0.25C, +0.50C, +0.75C, +1.0C, +1.25C, and +1.5C), or every ~15 minutes of (up to ~90 minutes) and immediately after heating
  Self-assessments of thermal comfort using four-point analog scale where 1 is "Not uncomfortable" and 4 is "Very uncomfortable"
Mental Acuity | For each study arm (all completed within 4 months), measurements taken 2 hours before heating (pre-pill ingestion), 5-minutes before initiating heating, and within 5-minutes after the heating protocol
  Indexed with digital Stroop test
Sleepiness/Fatigue level | For each study arm (all completed within 4 months), measurements taken 2 hours before heating (pre-pill ingestion), 5-minutes before initiating heating, and within 5-minutes after the heating protocol
  Measured using Stanford Sleepiness Scale (min: 1, max: 7 (more fatigued))

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University C.J Sanders Fieldhouse, Thunder Bay, Ontario, Canada